CLINICAL TRIAL: NCT05394857
Title: A Single-arm, Open-label, Prospective Phase II Study to Evaluate the Efficacy and Safety of SHR-1314 by Subcutaneous Injection in Active Moderate to Severe Graves' Orbitopathy Patients
Brief Title: Efficacy and Safety of SHR-1314 by Subcutaneous Injection in Active Moderate to Severe Graves' Orbitopathy Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor commercial considerations
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1314-205
Record Dates: First submitted 2022-05-23; First posted 2022-05-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Active Moderate to Severe Graves' Orbitopathy

STUDY DESIGN:
Intervention Model Description: SHR-1314 s.c in the treatment group, no placebo
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): SHR-1314 s.c
  Interventions: Drug: SHR-1314

INTERVENTIONS:
Drug: SHR-1314 — SHR-1314 subcutaneously

SUMMARY:
This is a single-arm, prospective, open-label, Phase II study that explored the efficacy and safety of SHR-1314 in active moderate to severe Graves' Orbitopathy. The study consists of a 6-week screening period, a 16-week treatment period, and a 12-week follow-up period. Eighteen adult patients with active moderate to severe Graves' Orbitopathy will be enrolled. Eligible subjects will receive SHR-1314 subcutaneously. The primary endpoint was the proptosis responder rate and will be evaluated at 16weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be able to understand and communicate with the investigator and comply with the requirements of the study and must give a written, signed and dated informed consent before any study assessment is performed.
2. Male or female between the ages of 18 and 70 (including boundary values)
3. Onset of active GO symptoms fewer than 9 months prior to baseline.
4. Clinical diagnosis of Graves' disease associated with active GO with a CAS ≥ 3 (on the 7-item scale) for the most severely affected eye(study eye) at Screening and Baseline.
5. Moderate-to-severe active GO (not sight-threatening but has an appreciable impact on daily life).
6. Does not require immediate surgical ophthalmological intervention.

Exclusion Criteria:

1. Pregnant or lactating women.
2. allergy to the study drug or to any component of the study drug.
3. Significant abnormalities in laboratory and ECG.
4. Decreased best corrected visual acuity due to optic neuropathy as defined by a decrease in vision of 2 lines on the Snellen chart, new visual field defect, or color defect secondary to optic nerve involvement within the last 6 months.
5. Corneal decompensation unresponsive to medical management.
6. Decrease in CAS of ≥ 2 points between Screening and Baseline.
7. Decrease in proptosis of ≥ 2 mm between Screening and Baseline.
8. Previous orbital irradiation or surgery for TED.
9. Any other ophthalmic disease that might interfere the study or the study result confirmed by investigator.
10. Patients with serious, progressive and uncontrolled cardiovascular, liver, kidney, lung, gastrointestinal, hematopoietic, endocrine, nervous and psychiatric diseases, or other conditions that considered inappropriate for patients to participate this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
the proptosis responder rate | week 16
  Proptosis responder is defined as a ≥ 2 mm reduction from Baseline in proptosis in the study eye, without deterioration [≥ 2 mm increase] of proptosis in the fellow eye)

SECONDARY OUTCOMES:
Proportion of patients achieving response in reduction of clinical activity score(CAS) | week 16
  reduction of CAS is defined as reduction of ≥ 2 points of CAS from Baseline to Week16.
Overall responder rate | week 16
  Overall responder rate is defined as percentage of subjects with≥ 2-point reduction in CAS AND ≥ 2 mm reduction in proptosis from Baseline, provided there is no corresponding deterioration [≥ 2-point/mm increase] in CAS or proptosis in the fellow eye at Week 16
The percentage of subjects with a CAS value of 0 or 1 in the study eye | week 16
  the clinical activity score of subject is 0 or 1.
The mean change from Baseline to Week 16 in proptosis measurement in the study eye | week 16
  Average change in proptosis in study eye.
Diplopia response rate at Week16 | week 16
  Proportion of participants with Baseline diplopia > 0 and a reduction of ≥ 1 grade with no corresponding deterioration (≥ 1 grade worsening) in the fellow eye at Week 16.
The mean change from Baseline to Week 16 in the GO-QoL score | week 16
  Average change in the Graves' ophthalmopathy quality of life questionnaire (GO-QOL) score. The GO-QoL contains 8 questions on visual functioning and 8 questions on appearance; answers on each subscale are transformed to scores ranging from 0 (worst) to 100 (best).

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Ninth People's Hospital,Shanghai Jiao Tong University School of Medical, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided